CLINICAL TRIAL: NCT07368192
Title: Community-Based Exercise Oncology: Real-World Evidence of High Adherence, Improved Quality of Life and Cost-Effectiveness Across the Cancer Continuum
Status: Active, not recruiting | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Universidad Pontificia Comillas (Other); Ejercicio y Cáncer (Community Exercise Program) (Unknown)
Responsible Party: Sponsor
Other Study IDs: COHORT-EYC-22-25
Record Dates: First submitted 2025-12-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Neoplams
Keywords: exercise oncology; Community-based program; Real-world evidence; Adherence; Quality of life; QALYs; Cost-effectiveness
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cancer survivors: Adults with a previous cancer diagnosis who had completed primary oncological treatment and were participating in a community-based supervised exercise oncology program.
- Active Cancer Treatment: Adults with a cancer diagnosis undergoing active oncological treatment, excluding hormonotherapy, who were participating in the supervised community-based exercise oncology program.
- Hormone therapy: Adults with a cancer diagnosis receiving hormonotherapy who were enrolled in the supervised community-based exercise oncology program.
- Metastatic: Adults with metastatic cancer participating in the supervised community-based exercise oncology program, with medical clearance for moderate-intensity exercise.

SUMMARY:
This prospective observational cohort study evaluates a community-based supervised exercise oncology program delivered in real-world settings in Madrid, Spain. The program is designed for adults with a cancer diagnosis across the cancer continuum, including survivors, patients undergoing active treatment, individuals receiving hormonotherapy, and patients with metastatic disease.

Participants take part in a structured multimodal exercise program combining aerobic, resistance, and functional training, delivered in supervised group-based sessions either in person or through synchronous online formats. The primary aims of the study are to assess program adherence, health-related quality of life, fatigue, and cost-effectiveness, expressed as quality-adjusted life years (QALYs). Secondary outcomes include cardiorespiratory fitness, muscular strength, functional capacity, physical activity levels, body composition, and psychological well-being.

Assessments are conducted at baseline and every four months over a 12-month follow-up period. This study provides real-world evidence on the feasibility, clinical impact, and economic value of community-based exercise oncology programs across different stages of the cancer trajectory.

DETAILED DESCRIPTION:
This study is a prospective observational cohort analysis of adults with a confirmed cancer diagnosis participating in a community-based supervised exercise oncology program in Madrid, Spain. Participants are referred by oncology specialists or self-referred with medical clearance to engage in moderate-intensity physical exercise.

The intervention consists of supervised multimodal exercise sessions lasting approximately 75 minutes, including warm-up, combined aerobic and resistance training, and cool-down periods. Aerobic training is prescribed using heart rate reserve and perceived exertion scales, while resistance training includes free-weight and functional exercises targeting major muscle groups. Sessions are delivered in small groups either face-to-face or via synchronous online platforms, with individualized progression and safety monitoring.

Participants undergo standardized assessments at baseline and at 4, 8, and 12 months. Primary outcomes include adherence to supervised exercise sessions, health-related quality of life, fatigue, and cost-effectiveness measured through quality-adjusted life years derived from EQ-5D instruments. Secondary outcomes include estimated cardiorespiratory fitness, muscular strength, functional capacity tests, physical activity behavior, body composition, and psychological outcomes.

The study aims to generate real-world evidence on the feasibility, effectiveness, and economic impact of integrating structured exercise programs into community-based cancer care across different clinical stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Confirmed diagnosis of cancer, at any stage of disease.
* Medical clearance to perform moderate-intensity physical exercise.
* Able to ambulate independently without assistive devices.
* Willingness to attend supervised exercise sessions for a follow-up period of at least 12 months.

Exclusion Criteria:

* Absolute medical contraindications to exercise (e.g., unstable angina, uncontrolled arrhythmias, severe anemia, acute infection, or thrombosis).
* Unstable metastatic bone disease without radiologic and/or oncologic clearance.
* Cognitive or functional impairment preventing safe participation in the exercise program.
* Concurrent participation in another structured exercise intervention or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults (≥18) with a confirmed cancer diagnosis.
  * At any stage of the disease.
  * Who have been medically cleared to participate in supervised exercise.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | Baseline, 4 months, 8 months, and 12 months.
  Percentage of supervised exercise sessions completed out of scheduled sessions.
Health-related quality of life (FACT-G) | Baseline, 4 months, 8 months, and 12 months.
  Health-related quality of life (units on a scale) assessed using the Functional Assessment of Cancer Therapy - General (FACT-G)
Fatigue (FACT-F) | Baseline, 4 months, 8 months, and 12 months.
  Fatigue (units on a scale) assessed using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACT-F).
Quality-adjusted life years (QALYs) | Baseline, 4 months, 8 months, and 12 months.
  Quality-adjusted life years calculated by integrating EQ-5D utility scores collected at multiple time points over the 12-month follow-up period. Repeated EQ-5D measurements are aggregated to derive a single QALY value per participant.
Barriers to participation | Baseline, 4 months, 8 months, and 12 months.
  Using a structured questionnaire based on previously published frameworks on determinants of adherence in cancer survivors.

SECONDARY OUTCOMES:
Estimated VO₂max | Baseline, 4 months, 8 months, and 12 months.
  Estimated maximal oxygen uptake (VO₂max) assessed using the Bruce treadmill protocol and Mackenzie equation.
Muscular strength | Baseline, 4 months, 8 months, and 12 months.
  Upper- and lower-limb muscular strength (kg) estimated using submaximal tests to estimate one-repetition maximum (1RM).
Functional capacity | Baseline, 4 months, 8 months, and 12 months.
  Functional capacity assessed using the 6-Minute Walk Test (6MWT) in meters.
Functional capacity | Baseline, 4 months, 8 months, and 12 months.
  Functional capacity assessed using the 30-second Sit-to-Stand test (repetitions)
Body weight (kg) | Baseline, 4 months, 8 months, and 12 months.
  Body weight assessed by bioelectrical impedance analysis using the Tanita MC-601F.
Body Fat Percentage (%) | Baseline, 4 months, 8 months, and 12 months.
  Body Fat Percentage (%) assessed by bioelectrical impedance analysis (Tanita MC-601F).
Fat Mass (kg) | Baseline, 4 months, 8 months, and 12 months.
  Fat Mass (kg) assessed by bioelectrical impedance analysis (Tanita MC-601F).
Lean Mass Percentage (%) | Baseline, 4 months, 8 months, and 12 months.
  Lean Mass Percentage (%) assessed by bioelectrical impedance analysis (Tanita MC-601F).
Lean Mass (kg) | Baseline, 4 months, 8 months, and 12 months.
  Lean Mass (kg) assessed by bioelectrical impedance analysis (Tanita MC-601F).
Physical activity | Baseline, 4 months, 8 months, and 12 months.
  Physical activity levels assessed using the International Physical Activity Questionnaire (IPAQ). The IPAQ estimates total physical activity expressed as metabolic equivalent minutes per week (MET-min/week), calculated from self-reported frequency, duration, and intensity of physical activity. Scores range from 0 MET-min/week to no upper limit, with higher values indicating higher levels of physical activity.
Anxiety (HADS-A) | Baseline, 4 months, 8 months, and 12 months.
  Symptoms of anxiety (units on a scale) assessed using the Hospital Anxiety Scale (HADS-A) The HADS-A consists of 7 items scored from 0 to 3, yielding a total score ranging from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
Depression (HADS-D) | Baseline, 4 months, 8 months, and 12 months.
  Depressive symptoms assessed using the Hospital Anxiety and Depression Scale - Depression subscale (HADS-D). The HADS-D consists of 7 items scored from 0 to 3, yielding a total score ranging from 0 to 21, with higher scores indicating greater severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Casla-Barrio, PhD., Principal Investigator — Director of the Exercise and Cancer Center
Locations (1):
- Ejercicio y Cáncer Center, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations, as the dataset includes sensitive health information collected in a real-world community-based program. Data are stored in accordance with local data protection regulations and institutional policies.

REFERENCES:
- [Result] Casla-Barrio S, Castellanos-Montealegre M, Pareja-Galeano H. The impact of multimodal high intensity exercise program comparing online and onsite interventions in breast cancer survivors: a randomized controlled trial. Clin Transl Oncol. 2026 Jan;28(1):184-192. doi: 10.1007/s12094-025-03979-x. Epub 2025 Jul 11. PMID 40643869
- See also: Official website of the community-based exercise oncology program where the supervised multimodal exercise intervention described in this study is delivered, including general information about the program structure and services. — https://ejercicioycancer.es/